CLINICAL TRIAL: NCT05710224
Title: A Phase 2, Randomized, Double-Blind, Multicenter, Safety and Immunogenicity Clinical Bridging Study to Compare V181 (Dengue Quadrivalent Vaccine rDENVΔ30 [Live, Attenuated]) to Butantan Dengue Vaccine (Butantan - DV) in Healthy Adults 18 to 50 Years of Age in Brazil
Brief Title: Clinical Bridging Study Between V181 (Dengue Quadrivalent Vaccine rDENVΔ30 [Live, Attenuated]) to Butantan Dengue Vaccine (Butantan - DV) in Healthy Adults 18 to 50 Years of Age in Brazil (V181 - 002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V181- 002; 25351.019896/2021- 84 (Other: Agência Nacional de Vigilância Sanitária (Brazilian Health Regulatory Agency) (ANVISA))
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- V181 (Experimental): Participants received a single 0.5 mL subcutaneous (SC) injection of V181.
  Interventions: Biological: V181
- Butantan - DV (Experimental): Participants received a single 0.5 mL SC injection of Butantan - DV.
  Interventions: Biological: Butantan - DV

INTERVENTIONS:
Biological: V181 — 0.5 mL SC dose of V181
  Arms: V181
Biological: Butantan - DV — 0.5 mL SC dose of Butantan - DV
  Arms: Butantan - DV

SUMMARY:
The purpose of this study was to demonstrate that V181 is safe and well tolerated and elicits an immune response that is non-inferior to that of Butantan - DV at Day 28 post-vaccination in adults 18 to 50 years of age in Brazil. The primary hypothesis was that V181 is non-inferior to Butantan - DV for each of the 4 dengue serotypes based on geometric mean titers (GMTs) and seroconversion rates at Day 28 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Male participants were eligible to participate if they agreed to the following for at least 90 days after administration of study intervention:

  * Abstained from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agreed to remain abstinent; or agreed to use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause).
* A female participant was eligible to participate if she was not pregnant or breastfeeding, and at least one of the following conditions applies:

  * was NOT a woman of child-bearing potential (WOCBP); or
  * was a WOCBP and using a contraceptive a highly effective method (with a failure rate of <1% per year), or
  * was abstinent from heterosexual intercourse as her preferred and usual lifestyle (abstinent on a long term and persistent basis), for at least 90 days after administration of study intervention.
  * Had a negative highly sensitive pregnancy test (urine or serum, as required by local regulations) before administration of study intervention
* Were dengue seronegative based on a pre-vaccination point of care (POC) dengue test.

Exclusion Criteria:

* Had a known history of dengue or Zika natural infection.
* Had an acute febrile illness (axillary temperature ≥37.8°C) occurring within 72 hours prior to receipt of study vaccine.
* Had a known hypersensitivity or history of severe allergic reaction (eg, swelling of the mouth and throat, difficulty breathing, hypotension or shock) to any component of the dengue vaccine, that required medical intervention.
* Had a serious or progressive disease, including but not limited to cancer, uncontrolled diabetes, severe cardiac, renal or hepatic insufficiency, systemic autoimmune or neurologic disorder.
* Had known or suspected impairment of immunological function, including but not limited to congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, hematologic malignancy, or treatment for autoimmune diseases.
* Had a condition in which repeated venipuncture or injections pose more than minimal risk, such as hemophilia, thrombocytopenia, other severe coagulation disorders, or significantly impaired venous access
* Had received a dose of any dengue vaccine (investigational or approved) prior to study entry or plans to receive any dengue vaccine (investigational or approved) for trial duration.
* Had received a licensed non-live vaccine within 14 days before receipt of study vaccine or was scheduled to receive any licensed non-live vaccine within 28 days following receipt of study vaccine. Exception: Inactivated influenza vaccine might be administered, but given at least 7 days before receipt of study vaccine or at least 28 days after receipt of study vaccine.
* Had received a licensed live vaccine within 28 days prior to receipt of study vaccine or was scheduled to receive any live vaccine within 28 days following receipt of study vaccine.
* Had received systemic corticosteroids (equivalent of ≥2 mg/kg/day of prednisone or ≥20 mg/day for persons weighing >10 kg) for ≥14 consecutive days and had not completed treatment at least 30 days before study entry or was expected to receive systemic corticosteroids at aforementioned dose and duration within 28 days following receipt of study vaccine. (Note: topical and inhaled/nebulized steroids were permitted.)
* Had received systemic corticosteroids exceeding physiologic replacement doses (approximately 5 mg/day prednisone equivalent) within 14 days before vaccination.
* Had received immunosuppressive therapies, including chemotherapeutic agents used to treat cancer or other conditions, treatments associated with organ or bone marrow transplantation, or autoimmune disease, within 6 months prior to receipt of study vaccine, or plans to receive immunosuppressive therapies within 28 days following receipt of study vaccine.
* Had received a blood transfusion or blood products (including immunoglobulins) within 6 months prior to receipt of study vaccine or plans to receive a blood transfusion or blood products (including immunoglobulins) within 28 days following receipt of study vaccine.
* Had planned donation of blood, eggs, or sperm at any time from signing the informed consent through 90 days post-vaccination.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1364 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Brazil (14):
  - Hospital Tacchini (Site 0006), Bento Gonçalves, Rio Grande do Sul
  - Fundação Universidade de Caxias do Sul (FUCS) - Instituto de Pesquisas em Saúde (IPS) (Site 0017), Caxias do Sul, Rio Grande do Sul
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia (Site 0005), Ijuí, Rio Grande do Sul
  - Hospital São Vicente de Paulo-Education and Research Management (Site 0007), Passo Fundo, Rio Grande do Sul
  - Instituto Méderi de Pesquisa e Saúde (0020), Passo Fundo, Rio Grande do Sul
  - Hospital Escola da Universidade Federal de Pelotas (Site 0009), Pelotas, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre-Centro de Pesquisa em Infectologia (Site # 003), Porto Alegre, Rio Grande do Sul
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul (Site 0011), Porto Alegre, Rio Grande do Sul
  - LMK Serviços Médicos S/S-Reumacenter (Site 0004), Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento - Centro de Pesquisa Clínica (Site0021), Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS-Centro de Pesquisa Clínica HSL-PUCRS (Site 0015), Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Santa Maria (UFSM) - Hospital Univer-Unidade de Pesquisa Clínica-UPC (Site 0001), Santa Maria, Rio Grande do Sul
  - Clínica Supera (Site 0019), Chapecó, Santa Catarina
  - Criciuma (Site 0008), Passo Fundo, Santa Catarina

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- V181: Participants received a single 0.5 mL subcutaneous (SC) injection of V181 .
- Butantan-DV: Participants received a single 0.5 mL SC injection of Butantan - DV.
Period: Overall Study
Arm/Group | V181 | Butantan-DV
Started | 682 | 682
Treated | 680 | 678
Completed | 660 | 665
Not Completed | 22 | 17
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 16 | 7
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Randomized By Mistake Without Study Treatment | 1 | 2
Not completed — Participants Left The City | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V181 | Butantan - DV | Total
Number analyzed (Participants) | 682 | 682 | 1364
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (8.9) | 32.2 (9.0) | 32.5 (9.0)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Male - participants with sex: male; Female - participants with sex: female; Undifferentiated - participant who is born with genitalia and/or secondary sexual characteristics of indeterminate sex, or which combine features of both sexes.
  Participants
    Male | 222 | 257 | 479
    Female | 459 | 425 | 884
    Undifferentiated | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 569 | 575 | 1144
  Not Hispanic or Latino | 99 | 92 | 191
  Unknown or Not Reported | 14 | 15 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 70 | 71 | 141
  White | 585 | 579 | 1164
  More than one race | 20 | 27 | 47
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dengue Virus (DENV)-Neutralizing Antibody Titers as Measured by Virus Reduction Neutralization Test (VRNT)
Description: A dengue VRNT was conducted to assess neutralizing antibody geometric mean titers (GMTs) for each of the 4 dengue serotypes (DENV1, DENV2, DENV3, and DENV4) in specimens collected from participants on Day 28 post-vaccination
Time Frame: Day 28 post-vaccination
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses and with data available for this outcome. These deviations included seropositivity at baseline as assessed by VRNT and missing serological results.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Butantan-DV: Participants received a single 0.5 mL SC injection of Butantan-DV.
Arm/Group | V181 | Butantan-DV
Number analyzed (Participants) | 514 | 531
Titer
  DENV-1 Serotype | 608.55 [550.54 to 672.66] | 703.19 [642.56 to 769.53]
  DENV-2 Serotype | 773.96 [711.16 to 842.30] | 109.05 [94.98 to 125.20]
  DENV-3 Serotype | 179.97 [161.27 to 200.83] | 396.76 [357.92 to 439.81]
  DENV-4 Serotype | 206.58 [180.71 to 236.16] | 593.41 [520.27 to 676.83]
Statistical Analysis 1: Comparison: V181 vs Butantan-DV; DENV-1 GMT Ratio (V181/Butantan - DV); Test type: Non-Inferiority — The statistical criterion for non-inferiority requires the lower bound of the 2-sided 95% CI for the GMT Ratio (V181 / Butantan - DV) to be >0.67; p < 0.001, t-distribution — p-value, GMT Ratio, and CI are calculated using t-distribution with the variance estimate from serotype specific linear model utilizing the natural log-transformed antibody titers as the response and a single term for vaccination group; GMT Ratio = 0.87, 95% CI 2-sided [0.76 to 0.99]
Statistical Analysis 2: Comparison: V181 vs Butantan-DV; DENV-2 GMT Ratio (V181 / Butantan - DV); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, t-distribution — p-value, GMT ratio, and CI are calculated using the t-distribution with the variance estimate from a serotype specific linear model utilizing the natural log-transformed antibody titers as the response and a single term for vaccination group; GMT Ratio = 7.10, 95% CI 2-sided [6.03 to 8.35]
Statistical Analysis 3: Comparison: V181 vs Butantan-DV; DENV-3 GMT Ratio (V181 / Butantan - DV); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 1.000, t- distribution — p-value, GMT ratio, and CI were calculated using the t-distribution with the variance estimate from a serotype specific linear model utilizing the natural log-transformed antibody titers as the response and a single term for vaccination group; GMT Ratio = 0.45, 95% CI 2-sided [0.39 to 0.53]
Statistical Analysis 4: Comparison: V181 vs Butantan-DV; DENV-4 GMT Ratio (V181 / Butantan - DV); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 1.000, t-distribution — [p-value comment as in outcome 1, analysis 3]; GMT Ratio = 0.35, 95% CI 2-sided [0.29 to 0.42]

2. Primary Outcome: Percentage of Participants Who Seroconverted, as Measured by VRNT
Description: A dengue VRNT was conducted to assess the percentage of participants who seroconverted for each of the 4 dengue serotypes (DENV-1, DENV-2, DENV-3 and DENV-4) at Day 28 post-vaccination. Seroconversion was defined as achieving a serotype-specific VRNT titer ≥lower limit of quantification (LLOQ) at Day 28 post-vaccination in the analysis population.
Time Frame: Day 28 post-vaccination
Population: All randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses and with data available for this outcome. These deviations included seropositivity at baseline as assessed by VRNT and missing serology results.
Measure: Number; unit: percentage of participants
Arm/Group | V181 | Butantan-DV
Number analyzed (Participants) | 514 | 531
percentage of participants
  DENV-1 Serotype | 98.6 | 98.9
  DENV-2 Serotype | 99.2 | 84.2
  DENV-3 Serotype | 95.3 | 98.9
  DENV-4 Serotype | 92.2 | 95.9
Statistical Analysis 1: Comparison: V181 vs Butantan-DV; DENV-1 Difference in percentage (V181 - Butantan-DV); Test type: Non-Inferiority — The statistical criterion for non-inferiority required the lower bound of the 2-sided 95% CI for the difference in percentages (V181 - Butantan-DV) to be >-10 percentage points; p < 0.001, Miettinen & Nurminen method — p-value, estimated difference in percentage, and CI were calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = -0.2, 95% CI 2-sided [-1.8 to 1.3]
Statistical Analysis 2: Comparison: V181 vs Butantan-DV; DENV-2 Difference in Percentage (V181 - Butantan-DV); Test type: Non-Inferiority — The statistical criterion for non-inferiority required the lower bound of the 2-sided 95% CI for the difference in percentages (V181 - Butantan - DV) to be >-10 percentage points; p < 0.001, Miettinen & Nurminen method — p-value, estimated difference in percentage, and CI were calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = 15.0, 95% CI 2-sided [12.0 to 18.5]
Statistical Analysis 3: Comparison: V181 vs Butantan-DV; DENV-3 Difference in Percentage (V181 - Butantan-DV); Test type: Non-Inferiority — The statistical criterion for non-inferiority requires the lower bound of the 2-sided 95% CI for the difference in percentages (V181 - Butantan-DV) to be >-10 percentage points; p < 0.001, Miettinen & Nurminen method — p-value, estimated difference in percentage, and CI are calculated using the unstratified Miettinen & Nurminen method; Difference in percentage = -3.5, 95% CI 2-sided [-5.8 to -1.6]
Statistical Analysis 4: Comparison: V181 vs Butantan-DV; DENV-4 Difference in Percentage (V181 - Butantan - DV); Test type: Non-Inferiority — The statistical criterion for non-inferiority requires the lower bound of the 2-sided 95% CI for the difference in percentages (V181 - Butantan - DV) to be >-10 percentage points; p < 0.001, Miettinen & Nurminen method — p-value, estimated difference in percentage, and CI are calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = -3.6, 95% CI 2-sided [-6.7 to -0.8]

3. Primary Outcome: Percentage of Participants With Vaccine-related Serious Adverse Events (SAEs)
Description: An SAE is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator.
Time Frame: Up to 28 days post-vaccination
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | V181 | Butantan-DV
Number analyzed (Participants) | 680 | 678
percentage of participants | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants Who Experience Solicited Injection-site Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs included erythema (redness), pain, and swelling.
Time Frame: Up to 5 days post-vaccination
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | V181 | Butantan-DV
Number analyzed (Participants) | 680 | 678
percentage of participants
  Injection-site erythema | 10.3 | 6.0
  Injection-site pain | 17.6 | 17.8
  Injection-site swelling | 2.8 | 2.2
Statistical Analysis 1: Comparison: V181 vs Butantan-DV; Erythema: Difference in Percentage (V181-Butantan - DV); Test type: Other — Estimated difference in percentage and CI were calculated using the unstratified Miettinen & Nurminen method; Difference in percentage = 4.2, 95% CI 2-sided [1.4 to 7.2]
Statistical Analysis 2: Comparison: V181 vs Butantan-DV; Pain: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI are calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = -0.2, 95% CI 2-sided [-4.3 to 3.9]
Statistical Analysis 3: Comparison: V181 vs Butantan-DV; Swelling: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI are calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = 0.6, 95% CI 2-sided [-1.1 to 2.3]

5. Secondary Outcome: Percentage of Participants Who Experience Solicited Systemic AEs
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs include arthralgia (joint pain), fatigue (tiredness), headache, myalgia (muscle pain), pyrexia (axillary temperature ≥37.8°C or 100°F), and rash.
Time Frame: Up to 28 days post-vaccination
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | V181 | Butantan-DV
Number analyzed (Participants) | 680 | 678
percentage of participants
  Arthralgia | 21.0 | 22.1
  Fatigue | 44.6 | 46.8
  Headache | 64.6 | 67.7
  Myalgia | 37.2 | 45.1
  Pyrexia | 5.6 | 10.8
  Rash | 70.6 | 63.7
Statistical Analysis 1: Comparison: V181 vs Butantan-DV; Arthralgia: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI were calculated using the unstratified Miettinen & Nurminen method; Difference in percentage = -1.1, 95% CI 2-sided [-5.5 to 3.3]
Statistical Analysis 2: Comparison: V181 vs Butantan-DV; Fatigue: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI are calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = -2.2, 95% CI 2-sided [-7.5 to 3.1]
Statistical Analysis 3: Comparison: V181 vs Butantan-DV; Headache: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI are calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = -3.1, 95% CI 2-sided [-8.2 to 1.9]
Statistical Analysis 4: Comparison: V181 vs Butantan-DV; Myalgia: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI were calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = -7.9, 95% CI 2-sided [-13.1 to -2.7]
Statistical Analysis 5: Comparison: V181 vs Butantan-DV; Pyrexia: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI are calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = -5.2, 95% CI 2-sided [-8.2 to -2.3]
Statistical Analysis 6: Comparison: V181 vs Butantan-DV; Rash: Difference in Percentage (V181 - Butantan - DV); Test type: Other — Estimated difference in percentage and CI were calculated using the unstratified Miettinen & Nurminen method; Difference in Percentage = 6.9, 95% CI 2-sided [1.9 to 11.8]

ADVERSE EVENTS:
Time Frame: Up to ~20 months
Description: All-cause mortality: All randomized participants; AEs: All randomized participants who received at least one dose of study intervention.
Groups:
- V181: Participants received a single 0.5 mL SC injection of V181.
Arm/Group | V181 | Butantan - DV
All-Cause Mortality (participants affected / at risk) | 1/682 | 0/682
Serious Adverse Events (participants affected / at risk) | 12/680 | 9/678
Other Adverse Events (participants affected / at risk) | 634/680 | 622/678
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V181 (N=680) | Butantan - DV (N=678)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis A (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V181 (N=680) | Butantan - DV (N=678)
Eye Pain (Eye disorders) | 32 (32) | 40 (42)
Nausea (Gastrointestinal disorders) | 41 (43) | 36 (38)
Fatigue (General disorders) | 294 (294) | 311 (312)
Injection site erythema (General disorders) | 72 (72) | 45 (45)
Injection site pain (General disorders) | 121 (121) | 124 (124)
Pyrexia (General disorders) | 46 (49) | 92 (101)
Arthralgia (Musculoskeletal and connective tissue disorders) | 139 (141) | 147 (149)
Pruritus (Skin and subcutaneous tissue disorders) | 57 (57) | 67 (70)
Rash (Skin and subcutaneous tissue disorders) | 480 (482) | 432 (435)
Myalgia (Musculoskeletal and connective tissue disorders) | 242 (242) | 294 (297)
Headache (Nervous system disorders) | 421 (429) | 441 (443)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor and Merck Sharp & Dohme LLC (MSD), the investigator agrees to submit all manuscripts or abstracts to the Sponsor and MSD before submission. This allows the Sponsor and MSD to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT05710224/Prot_SAP_000.pdf